CLINICAL TRIAL: NCT00069849
Title: A Study of the Safety and Efficacy of Multiple Doses of ABT-089 in Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M03-614
Record Dates: First submitted 2003-10-01; First posted 2003-10-02 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — pozanicline

INTERVENTIONS:
Drug: ABT-089

SUMMARY:
The purpose of this study is to compare the safety and efficacy of 2 mg, 4 mg, and 20 mg of ABT-089 BID to placebo in adults with Alzheimer's disease.

ELIGIBILITY:
INCLUSION CRITERIA:

* Current diagnosis of probable Alzheimer's disease.
* ADAS-cog score of at least 12 and MMSE score of 10 to 26.
* Non-smoker
* Must have legally authorized representative and a reliable caregiver. The caregiver and legally authorized representative may be the same person.
* Fluent in English.

EXCLUSION CRITERIA:

* Use of cholinesterase inhibitors or any other drugs to treat Alzheimer's disease in the last 6 weeks.
* Has clinically significant or uncontrolled medical condition other than Alzheimer's disease.
* Nursing home resident.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2003-07

PRIMARY OUTCOMES:
MMSE

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Tracy, M.D., Study Director — Abbott
Locations (8):
- United States (8):
  - Fresno, California
  - San Diego, California
  - Orlando, Florida
  - West Palm Beach, Florida
  - Florence, Kentucky
  - Portland, Oregon
  - Salt Lake City, Utah
  - Bennington, Vermont